CLINICAL TRIAL: NCT03776474
Title: Determine Immunoglobulin G4 (IgG4) Standards for Cow's Milk and Egg in Different Populations of Allergic and Non-allergic Children
Acronym: IgG4
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180057; 2018-A01972-53 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-12-06; First posted 2018-12-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Food Allergy in Children
Keywords: Food allergy in children; Immunoglobulin E; Immunoglobulin G4; Oral food challenge; Plasma metabolomic analysis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Allergic: Minors allergic to cow's milk and/or eggs
  Interventions: Biological: Blood collection
- Non-allergic: Minors without history of allergy to cow's milk and/or eggs
  Interventions: Biological: Blood collection
- Acquired tolerance: Minors formerly allergic to cow's milk and/or eggs
  Interventions: Biological: Blood collection

INTERVENTIONS:
Biological: Blood collection — Patients less than 5 kg : 2 ml Patients over 5 kg : 3 ml Patients over 10 kg : 5 ml

SUMMARY:
The study objectives are :

Determine standards of plasma levels of casein-specific immunoglobulin G4 (IgG4) and egg-specific immunoglobulin G4 (IgG4) as a function of age, in non-allergic children, in allergic children, and in cured former allergic patients.

Analyze the plasma IgG4 / IgE ratio, according to the result of the oral provocation test (tolerance versus allergy) and, in the event of a reaction, according to the reactogenic dose (dose which caused the reaction).Determine whether analysis of the plasma metabolome can identify children with a cured allergy to cow's milk protein or to egg from those with a persistent allergy.

DETAILED DESCRIPTION:
Immunoglobulin E (IgE) mediated allergies to cow's milk and hen's egg affects 2-3% and 0.5-2.5% of children respectively. These allergies expose to the risk of immediate anaphylactic reaction that may be life-threatening. Approximately 70-80% of children with IgE mediated allergies to cow's milk and hen's egg will tolerate these foods by the age of 6 years. However, in the absence of reliable biomarker of tolerance, to determine whether oral tolerance is obtained, it is recommended to perform an oral food challenge (OFC) in a hospital setting. This procedure is expensive, time consuming, and carries the risk of anaphylactic reactions. Many studies have tried to find predictive markers of reactivity during the OFC. Improving the prediction of the response to OFC would be very useful to better select children in whom an OFC can be performed without risk to confirm the acquisition of tolerance.

For instance, serum specific IgE positive values beyond which 95% of patients would have an allergic reaction have been proposed. These values are highly variable from one study to another because of methodological differences and heterogeneity of populations, and cannot be used in clinical practice.

The regular dosage of serum specific IgE and its evolution over time is used in clinical practice to predict a possible persistence of IgE mediated food allergy. Indeed, an initial high rate and/or elevation of specific IgE levels may be predictive of a persistent allergy, while initial low rates and a decrease in specific IgE may predict tolerance. When tolerance develops, there is a decrease in specific IgE levels, however, even if tolerance is obtained, they can remain positive at pathological levels.

During continuous exposure to an allergen, the specific immunoglobulin G4 (IgG4) response is physiological. Oral immunotherapy studies in food allergies showed an elevation of specific IgG4, associated with an elevation in the number of regulatory T lymphocytes (LTreg) and the production of interleukin (IL)-10. The development of spontaneous oral tolerance, without the intervention of immunotherapy, also seems to involve IgG4. In a prospective follow-up of a cohort of children with an IgE-mediated cow's milk allergy, the elevation of specific IgG4 was observed in those who cure of their allergy, with rates higher than those observed in children whose allergy persists. In children with cow's milk and/or egg allergies, a low concentration of specific (IgG4 of B-Lactoglobulin or ovalbumin is associated with the need for a more prolonged exclusion diet. The balance between specific IgE and IgG4 therefore appears to be important in the development of tolerance and may reflect the balance between effector T cells and LTreg. However, the normal serum levels of IgG4 to cow's milk and hen's egg are unknown.

A recently published study of Doctor Guillaume Lezmi and Professor Karine Adel-Patient shows that children with an IgE-mediated allergy to cow's milk protein and those who outgrew this allergy, have distinct plasma metabolomic signature. This suggests that plasma metabolomic analysis may be a useful too to differentiate children with a persistent cow's milk protein allergy from those who acquired tolerance to cow's milk. If confirmed, the metabolic signature may be useful to better identify children to whom an oral food challenge with cow's milk protein could be propose. These results need to be confirmed in a larger population and in other food allergies.

The study objectives are :

Determine standards of plasma levels of casein-specific immunoglobulin G4 (IgG4) and egg-specific immunoglobulin G4 (IgG4) as a function of age, in non-allergic children, in allergic children, and in cured former allergic patients.

Analyze the plasma IgG4 / IgE ratio, according to the result of the oral provocation test (tolerance versus allergy) and, in the event of a reaction, according to the reactogenic dose (dose which caused the reaction).

Determine whether analysis of the plasma metabolome can identify children with a cured allergy to cow's milk protein or to egg from those with a persistent allergy.

ELIGIBILITY:
Inclusion Criteria:

* Minors aged 0 to 18
* In consultation or hospitalized for an oral food challenge for milk or eggs
* To undergo a blood test

Exclusion Criteria:

Minors with immune deficiency, chronic inflammatory disease or immunosuppressive or immunomodulator treatment

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Minors in consultation or hospitalized at Necker Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2025-11-18 (Estimated); Study Completion 2025-11-18 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of casein-specific immunoglobulin G4 and egg-specific immunoglobulin G4 | Day 0

SECONDARY OUTCOMES:
Plasma concentration of casein-specific immunoglobulin E and egg-specific immunoglobulin E | Day 0
Total immunoglobulin E plasma concentration | Day 0
Plasma concentration of casein-specific immunoglobulin G4 / plasma concentration of casein-specific immunoglobulin E ratio | Day 0
Plasma concentration of egg-specific immunoglobulin G4 / plasma concentration of egg-specific immunoglobulin E ratio | Day 0
Plasma concentration of casein-specific immunoglobulin G4 / total immunoglobulin E plasma concentration ratio | Day 0
Plasma concentration of egg-specific immunoglobulin G4 / total immunoglobulin E plasma concentration ratio | Day 0
Plasma metabolomic analysis | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Lezmi, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adel-Patient K, Lezmi G, Castelli FA, Blanc S, Bernard H, Soulaines P, Dumond P, Ah-Leung S, Lageix F, de Boissieu D, Cortes-Perez N, Hazebrouck S, Fenaille F, Junot C, Dupont C. Deep analysis of immune response and metabolic signature in children with food protein induced enterocolitis to cow's milk. Clin Transl Allergy. 2018 Sep 28;8:38. doi: 10.1186/s13601-018-0224-9. eCollection 2018. PMID 30275944